CLINICAL TRIAL: NCT04060121
Title: Efficacy of Psychological Therapies in Patients With Functional Bowel Disorders With History of Early Adverse Life Events or Post-traumatic Stress Disorder
Brief Title: Efficacy of Psychological Therapies in Patients With Functional Bowel Disorders
Acronym: PTSD
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other); Indiana Clinical and Translational Sciences Institute (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Huiping Xu, Associate Professor, Indiana University
Other Study IDs: 1802270023; UL1TR002529 (NIH)
Record Dates: First submitted 2019-08-13; First posted 2019-08-16 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: IBS - Irritable Bowel Syndrome; Constipation
Keywords: early adverse life events; ptsd; cognitive behavioral therapy
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is study bowel symptoms, quality of life, and personal factors that may affect your health. In Aim 1 of this study participants will be invited to complete 6 survey-based questionnaires online.

In Aim 2 of this study will monitor the effectiveness of a 12 week therapy program on bowel symptoms and overall quality of life.

DETAILED DESCRIPTION:
For Aim 1, investigators will conduct a cross-sectional survey study examining prevalence of early adverse life events and post-traumatic stress disorder (PTSD) in patients with constipation-predominant IBS or chronic constipation with or without overlapping dyssynergic defecation.

For Aim 2, investigators will recruit and enroll individuals who have a positive history of early adverse life events or possible PTSD as identified in Aim 1 for a 12 week outpatient cognitive behavioral therapy program as outlined below:

Visit 1 (Participants will present to the GI Office at one of our dedicated locations including the downtown Digestive and Liver Disorders (DaLD) clinic, Springmill Clinic, or IU North Multispeciality Clinic) At this screening visit, participants do the following:

* Read and sign the informed consent after all your questions about the study will be answered
* Have a medical history taken including demographics, symptoms and history of illness
* Medications will be reviewed
* A physical exam will be performed by the physician if the visit is being conducted in person. If the visit is done virtually, the physician will record that exam as a virtual exam with all relevant information that can be gathered by a virtual exam.
* Vital signs will be measured if the visit is conducted in person. If the visit is virtual, vital signs will not be physically done but any available data pertaining to vital signs will be documented.
* Participants will be asked to complete a series of questionnaires
* Participants will be provided a bowel pattern diary to record bowel symptoms over the course of the study
* Participants will be asked to complete global assessment scales (2 questions) during each week of the study
* Participants will be administered the PAC-SYM, PAC-QOL, global assessment scale, SF-12, HADS and PCL-5 during CBT
* Participants will be administered the GAD-7 and PHQ-9 at every CBT visit.
* The study visit may take 30 minutes to 1 hour to complete

Day 1-15 (Run-In Phase):

• Participants be asked to record stool symptoms and patterns in a diary daily starting from Day 1 to Day 15. The daily dairy can either be completed on paper or by phone or on the web.

Day 16-100 (Visit 2-13): During this time, participants will undergo regular sessions with a dedicated GI psychologist. They will receive one 60-minute session every week for 10-12 weeks. The treatment schedule will include education on the relationship between bowel symptoms and stressful life events with instructions on ways to cope and manage symptoms through the use of relaxation techniques, such as breathing exercises and other methods for self calming. During the 10 to 12 weeks of therapy, participants will be given assignments and asked to monitor your progress. After you have completed your treatment sessions, you will be asked to fill out the same questionnaires that you completed at your screening visit that can be done either in person using a physical form or virtually online.

Visit 14:

• We will also confirm completion of the study.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

-Patients with a history of constipation based on clinical evaluation undergoing diagnostic testing for dyssynergic defecation with anorectal manometry with balloon expulsion test, ages 18 years or older.

Aim 2:

* Patients with a history of constipation with or without dyssernergic defecation and a positive history of EALs or PTSD, as identified in Aim 1 based on survey responses.
* Any positive history regardless of symptom severity will be considered. Positive history will be defined by an ACE score of 1 or higher OR a provisional diagnosis of PTSD. A provisional PTSD diagnosis can be made by treating each PCL-5 item rated as 2 = "Moderately" or higher as a symptom endorsed. The diagnostic rule will require a rating of "moderate" for the following: 1 B item (questions 1-5), 1 C item (questions 6-7), 2 D items (questions 8-14), and 2 E items (questions 15-20).

Exclusion Criteria:

For Aim 1, key exclusion criteria are:

* Patients who are currently hospitalized
* Patients who are unable to consent
* Patients with microscopic colitis, inflammatory bowel disease, or celiac disease, visceral cancer, or uncontrolled thyroid disease.

In Aim 2, key exclusion criteria will include the aforementioned criteria listed in Aim 1 as well as the following:

* Patients who have bipolar disorder including active or recent hypomanic/manic episode
* Patients at imminent risk for harm to self or others
* Patients unable to follow orders
* Patients who have a history of organic brain disease
* Patient using illicit substances
* Pregnant or post-partum patients
* Patients who are homeless or lacking sufficient social support for follow-up care
* Patients with acute stress disorder as determined by the GI psychologist
* Patients with or severe PTSD as determined by the GI psychologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults' ages 18 years or older will be eligible for participation. We will solicit participation and extend survey invitations to participants who have undergone clinical evaluation for constipation with anorectal manometry and balloon expulsion testing at the IU GI Motility Laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Early adverse life events (EALS) | 10-15 minutes
  Presence of early adverse life events will be determine by self-reported questionnaire responses to the adverse childhood experiences (ACE) questionnaire (ACE score of one or higher, range 0-8)
Post-traumatic Stress Disorder (PTSD) | 10-15 minutes
  Prevalence of PTSD will be determined by self-reported questionnaire responses to PTSD Checklist (PCL-5) questionnaire (range 0-80). A provisional PTSD diagnosis can be made by treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 B item (questions 1-5), 1 C item (questions 6-7), 2 D items (questions 8-14), 2 E items (questions 15-20).
Change in weekly number of complete spontaneous bowel movements | 12 weeks
  The weekly number of complete spontaneous bowel movements will be measured using a validated daily bowel diary
Change in abdominal pain | 12 weeks
  Abdominal pain will be measured using a validated daily bowel diary

SECONDARY OUTCOMES:
IBS or functional constipation (FC) | 20-30 minutes
  Presence of IBS or FC will be determined based on responses to the validated IBS Rome IV Questionnaire
Psychological comorbidities | 20-30 minutes
  Existence and severity of psychological comorbidities will be measured by the validated hospital anxiety and depression scale (HADS) questionnaire (range 0-14)
Health-related quality of life: Short Form-12 (SF-12) | 20-30 minutes
  Health-related quality of life will be measured by responses to SF-12 (higher score is better, range 0-100)
Constipation-related symptoms | 12 weeks
  Change in constipation-related symptoms will be measured using the validated in Patient Assessment of Constipation Symptoms questionnaire (higher score is worse, score range 0-4)
Constipation-related quality of life | 12 weeks
  Change in constipation-related quality of life will be measured using the validated patient assessement of constipation quality of life questionnaire (higher score is worse, score range 0-4)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of medicine, Indianapolis, Indiana, United States